CLINICAL TRIAL: NCT06661993
Title: Effect of Alpha-lipoic Acid in Critically Ill Patients With Sepsis
Brief Title: Alpha-lipoic Acid in Critically Ill Patients With Sepsis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damanhour University (Other)
Collaborators: Tanta University (Other)
Responsible Party: Principal Investigator, Rehab Werida, Associate Professor, Damanhour University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: alpha-lipoic acid in sepsis
Record Dates: First submitted 2024-10-25; First posted 2024-10-28 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis | interventions — Thioctic Acid

STUDY DESIGN:
Intervention Model Description: 80 septic patients will be enrolled from Damanhur National medical institute, and they will be randomized using simple randomization into two groups (40 patients each): control group will receive placebo and ALA group will be given 1800 mg orally or via a nasogastric tube of ALA daily for seven days .
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Group (Placebo Comparator): control group: 40 septic patients will receive placebo daily for seven days.
  Interventions: Other: Placebo
- ALA group (Active Comparator): ALA group: 40 septic patients will be given 1800 mg orally or via a nasogastric tube daily for seven days .
  Interventions: Dietary Supplement: Alpha-lipoic acid

INTERVENTIONS:
Other: Placebo — placebo film-coated tablet orally or via a nasogastric tube for seven days .
  Other Names: placebo film-coated tablet
  Arms: Placebo Group
Dietary Supplement: Alpha-lipoic acid — Alpha-lipoic acid 1800 mg orally or via a nasogastric tube for seven days .
  Other Names: Thiotacid 1800 mg
  Arms: ALA group

SUMMARY:
Evaluate the of effect of alpha-lipoic acid in critically ill septic patients. 80 septic patients will be enrolled from Damanhur National medical institute, and they will be randomized using simple randomization into control group will receive placebo and ALA group will be given 1800 mg orally or via a nasogastric tube of ALA daily for seven days .

DETAILED DESCRIPTION:
1. Ethical committee approval will be obtained from ethics committee of Faculty of Pharmacy, Damanhour University & Ethics committee of Damanhur National Medical National Institute.
2. All participants or their relatives should agree to take part in this clinical study and will provide informed consent.
3. 80 septic patients will be enrolled from Damanhur National medical institute, and they will be randomized using simple randomization into control group will receive placebo and ALA group will be given 1800 mg orally or via a nasogastric tube of ALA daily for seven days .
4. Statistical tests appropriate to the study design will be conducted to evaluate the significance of the results.
5. Results, conclusion, discussion and recommendations will be given. Outcomes 1. The primary outcome ICU and hospital mortality, ICU and hospital stay, new acute kidney injury in ICU, demand and duration of life support, Sequential Organ Failure Assessment (SOFA)/Acute Physiology and Chronic Health Evaluation II (APACHE II) 2. The secondary outcome are as follows: A. 28-day all-cause mortality B. change in inflammatory markers such as CRP , IL6, and TNF Alpha and may be measured glycocalyx degradation markers such as syndecan 1.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will be diagnosed with sepsis or develop sepsis during their ICU length of stay
* Age 18 year and older
* Patient able to receive oral or enteral medication

Exclusion Criteria:

* Patients who will be diagnosed with septic shock
* Female patients who are pregnant or lactating.
* Participation in another clinical trial.
* Current treatment with other medications that have antioxidant effects, such as vitamin C and vitamin E.
* Allergy to LA or similar active agents (e.g., vitamin B), or previous intolerance to the recommended dose of LA

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-10-28 (Actual); Study Completion 2025-10-28 (Actual)

PRIMARY OUTCOMES:
Sequential Organ Failure Assessment (SOFA) Score | 1 week
  The SOFA score is a composite score based on the degree of dysfunction in six organ systems-respiratory, coagulation, hepatic, cardiovascular, central nervous system, and renal. Each organ dysfunction scores from 0 to 4, with increasing scores reflecting more abnormal physiology and biochemistry or an increasing degree of intervention. The higher the SOFA score, the higher the likely mortality.
ICU and hospital stay | 1 month
  Duration (days)

SECONDARY OUTCOMES:
Syndecan 1 (ug/dl) | 1 Week
  glycocalyx degradation marker
CRP (ug/dl) | 1 Week
  Inflammatory marker

CONTACTS AND LOCATIONS:
Overall Officials: Tarek Mostafa, Prof., Study Chair — Tanta University
Locations (1):
- Damanhour Teaching Hospital, General Organization for Teaching Hospitals and Institutes., Damanhūr, Elbehairah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rahimlou M, Asadi M, Banaei Jahromi N, Mansoori A. Alpha-lipoic acid (ALA) supplementation effect on glycemic and inflammatory biomarkers: A Systematic Review and meta- analysis. Clin Nutr ESPEN. 2019 Aug;32:16-28. doi: 10.1016/j.clnesp.2019.03.015. Epub 2019 May 2. PMID 31221283
- [Background] Thompson K, Venkatesh B, Finfer S. Sepsis and septic shock: current approaches to management. Intern Med J. 2019 Feb;49(2):160-170. doi: 10.1111/imj.14199. PMID 30754087